CLINICAL TRIAL: NCT03266939
Title: Rebalancing the Serotonergic System in Cocaine Dependence
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never funded because lorcaserin was pulled from FDA approval
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Amy C. Janes, Principal Investigator, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: cocaine and serotonin
Record Dates: First submitted 2017-08-23; First posted 2017-08-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet
- Active Medication (Active Comparator)
  Interventions: Drug: Lorcaserin

INTERVENTIONS:
Drug: Lorcaserin — 10 mg acute administration of lorcasein
  Arms: Active Medication
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo

SUMMARY:
In the United States, 1.5 million people abuse cocaine leading to a host of negative health and economic consequences, yet no FDA approved treatment exists. To develop effective treatments, the following must be considered: 1) do potential medications ameliorate brain disruptions associated with cocaine use? 2) are multiple, targeted treatments necessary? To meet these goals, innovative multi-modal neuroimaging will be used to determine whether rebalancing the serotonergic (5-HT) system reduces cocaine cue reactivity, impulsivity, and normalizes related neurochemistry and brain connectivity.

ELIGIBILITY:
Inclusion Criteria:

* - Participants will be male and female volunteers between the ages of 18-55
* Participants will report having used cocaine on at least four occasions within the month prior to screening; the urine sample obtained during the screening visit must be positive for the cocaine metabolite benzoylecgonine (>300 ng/ml). They can meet DSM-IV criteria for cocaine abuse and dependence.
* Participants cannot meet DSM-IV criteria for current psychotic disorders (e.g., bipolar disorder, schizophrenia, schizoaffective disorder)
* Participants cannot meet DSM-IV criteria for a current major depressive episode
* Participants cannot meet DSM-IV criteria for current drug dependence (except nicotine, cocaine, and marihuana)
* Participants must test negative for alcohol use on the day of the scan.
* Participants can report current abuse of marihuana and tobacco. Participants cannot have used marihuana within twelve hours of their study visits.
* Participants cannot be regular opiate users including prescription opiate analgesics
* Participants cannot have a history of major head trauma resulting in cognitive impairment, seizure, or other neurological disorders.
* Participants cannot have any conditions that are contraindicated for MRI (see next section)
* Participants cannot be pregnant (pregnancy test will be performed before each scanning session)
* Participants must be able to read screening materials including consent form and give informed consent
* Participants cannot be taking any medications with a 5-HT mechanism including serotonin-norepinephrine reuptake inhibitors (SNRIs), selective serotonin reuptake inhibitors (SSRIs), tricyclic antidepressants (TCAs), monoamine oxidase inhibitors (MAOIs) and St. John's Wort and tryptophan.
* Participants cannot be currently taking any medications that might affect the central nervous system including prescription analgesics, anxiolytics, antipsychotics, and antidepressants. A complete review of medications will be evaluated by study staff.
* Cannot have any history of a medical condition that might affect the central nervous system at the time of scanning including: Abnormal structural MRI, or a history of head trauma or injury causing loss of consciousness lasting longer than 3 minutes or associated with skull fracture or intracranial bleeding or who had irremovable magnetically active objects on or within their body, or history of epilepsy.

Exclusion Criteria:

* - Weight greater than 350 pounds (cannot easily fit inside the magnet bore)
* Cardiac pacemakers
* Aneurysm clips and other vascular stents, filters, clips or other devices
* Prosthetic heart valves
* Other prostheses
* Neuro-stimulator devices
* Implanted infusion pumps
* Cochlear implants
* Ocular implants or known metal fragments in eyes
* Exposure to shrapnel or metal filings (sheet metal workers, welders, and others)
* Other metallic surgical hardware in vital areas
* History of major head trauma resulting in cognitive impairment
* Certain tattoos (e.g. older dye with metallic pigment)
* Certain medication patches (if they cannot be removed)
* Metal containing IUDs
* Claustrophobia
* Pregnancy
* Metallic implants except fillings and crowns
* Tattoos containing metallic ink on the neck, shoulders, upper arm, and head (these could become heated during scanning, potentially causing burns
* Medication patches that cannot be removed during scanning
* Claustrophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Influence of lorcaserin on fMRI measured brain-reactivity to drug cues. | fMRI measures will be gathered on scanning visits 1 and 2 (approx 1 week apart)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Janes, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No